CLINICAL TRIAL: NCT05962437
Title: Three-arm Randomized Controlled Trial Investigating the Effectiveness, Cost-utility, and Physiological Effects of the Spanish Version of STANZA®: A Self-guided Digital Acceptance and Commitment Therapy (ACT) for Fibromyalgia
Brief Title: Self-guided Acceptance and Commitment Therapy-based Digital Smartphone Application for Management of Fibromyalgia
Acronym: SMART-FM-SP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Swing Therapeutics, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PI22/00829
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- STANZA-Spain (Experimental): Digital Acceptance and Commitment Terapy (ACT). It consists of 41 structured ACT lessons, incorporating mindfulness practices and daily activities to facilitate behavior change and promote gradual pacing of daily activities and exercise. The core content was designed to be completed within 8 weeks, with a 4-week maintenance period thereafter to strengthen skills.
  Interventions: Device: Self-guided digital Acceptance and Commitment Therapy; Behavioral: Treatment as Usual (TAU)
- FibroST-Spain (Active Comparator): A digital active control intervention is implemented to control for study engagement, expectations, and healthcare provider interaction biases. Components of this active comparator include daily symptom and function tracking (Daily Symptom Tracker), symptom and function monitoring, and access to health education articles about fibromyalgia.
  Interventions: Device: FM symptom tracking app (FM-ST); Behavioral: Treatment as Usual (TAU)
- Treatment as Usual (TAU) (Active Comparator): Usual care is mainly carried out by general practitioners and rheumatologists through regular consultations. Clinicians prescribe medications and provide some counselling.
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Device: Self-guided digital Acceptance and Commitment Therapy — Smartphone-based mobile health application (app) that delivers a self-guided, evidence-based ACT program tailored to the management of FM. This investigational digital therapeutic, referred to herein as STANZA, was inspired by a web-based ACT program for FM validated by University of Manitoba and was recently granted De Novo clearance by the U.S. FDA. The app delivers ACT in 15- to 20-minute daily doses over the course of 12 weeks without the involvement of healthcare providers. The program consists of interactive educational materials that teach ACT skills which are reinforced experientially via values exploration and identification, mindfulness, and relaxation exercises. Values-based assignments follow each lesson to assist patients in incorporating ACT skills into their daily lives. Uniquely, STANZA teaches additional skills, including self-guided physical exercise and pacing daily activities via a personally customized stepwise, gradual approach.
  Arms: STANZA-Spain
Device: FM symptom tracking app (FM-ST) — Based on the same platform as STANZA, FM-ST enables self-guided daily tracking of patient-reported symptoms and functioning. Symptom tracking is commonly used in chronic pain management. FM-ST also provides access to educational materials relevant to FM and general health but does not provide any psychotherapy or healthcare professional involvement. This app mitigates potential expectation, treatment time and attention, and healthcare provider interaction biases that often occur in chronic pain studies that utilize passive comparison conditions.
  Arms: FibroST-Spain
Behavioral: Treatment as Usual (TAU) — Usual care is mainly carried out by general practitioners and specialists in regular consultations, commonly consisting of face-to-face visits to monitor the physical and emotional status of the patient. Clinicians usually provide advice about physical exercise, diet, etc., and prescribe pharmacotherapy (pain medications, hypnotics and antidepressants)

SUMMARY:
Introduction: Fibromyalgia (FM) is a prevalent syndrome that lacks curative treatment, imposing high healthcare and societal costs. The SMART-FM-Spain study investigates the effectiveness, physiological effects, and cost-utility of a self-guided digital intervention (STANZA-Spain) based on Acceptance and Commitment Therapy (ACT) for patients with FM.

Methodology: Six-month, 3-arm randomized controlled trial (RCT) A total of 360 adult individuals meeting the 2016 American College of Rheumatology (ACR) criteria for FM will be recruited mainly at Vall d'Hebron University Hospital (Barcelona, Spain), and will be randomly allocated to one of the three study arms: Treatment as usual (TAU) plus STANZA-Spain, TAU plus digital symptom tracking (FibroST), or TAU. Participants will be assessed at baseline, post-treatment, and 6 month-follow-up. The primary outcome will be functional impairment and secondary outcomes will include patient impression of change, depression-anxiety-stress, and pain catastrophizing, among others constructs relevant to FM. Effectiveness and cost-utility analysis from a societal perspective will be computed, whereas ACT-related constructs, such as psychological flexibility, will be assessed to identify processes of change that will be analyzed with path analyses. Biomarkers will be assessed at baseline and post-treatment including hair cortisol, cortisone, corticosteroid binding globulin (CBG), adrenocorticotropic hormone (ACTH), cortisol in plasma, genotyping of FKBP5 gene polymorphisms, immune-inflammatory markers, and vitamin D levels.

Discussion: This study might represent a significant advancement in the management of FM in Spanish-speaking patients with FM, by examining the effectiveness, physiological effects, and cost-utility of a smartphone-based digital therapeutic with demonstrated empirical support in the United States of America.

DETAILED DESCRIPTION:
Main goals of the SMART-FM-SP study The main objectives of this RCT are: To analyze the effectiveness of adding Acceptance and Commitment Therapy via app (STANZA) compared to an active control arm (Fibro Symptom Tracker app -FibroST-) to the treatment as usual (TAU) for patients diagnosed of fibromyalgia; To examine the cost-utility of STANZA from healthcare and societal perspectives; To measure a set of biomarkers alongide the RCT in order to know the physiological underpinnings of the digital intervention STANZA and to identify potential predictors of treatment response.

Smart-FM-SP is a 6-months RCT with three arms: TAU, TAU+STANZA and TAU+FibroST. Therefore, patients in three arms will receive TAU, and FibroACT and FibroST will be complementary treatments to the standard one provided in the public Catalan Health System.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia diagnosis according to the 2016 ACR criteria
* Fibromyalgia Impact Questionnaire Revised (FIQR) total score within the range of 35-80 at baseline.
* Willing to maintain their current pain treatment throughout the study.
* Having a smartphone (iOS 12 or higher or Android OS 8 or higher).
* Proficient understanding of Spanish.

Exclusion Criteria:

* Presence of cognitive impairment according to clinical records.
* Diagnosis of severe medical or mental disorders such as cancer, psychotic disorder, and drug abuse according to medical records.
* Patients at risk of suicide.
* Being pregnant or planning a pregnancy during the study period, or currently breastfeeding.
* Participation in other clinical trials during the study or within the previous 90 days.
* Unable to use a smartphone.

Exclusion criteria for biomarkers substudy (50% of patients in each study arm):

* Comorbid rheumatologic disorders such as lupus.
* History of fever (> 38ºC), or infection within the last 2 weeks.
* Recent vaccination within the last 4 weeks.
* Needle phobia.
* Consumption of more than 8 units of caffeine per day.
* Smoking more than 5 cigarettes per day.
* Having hair length less than 3 cm.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire Revised (FIQR) | Through study completion, an average of 6 months
  The FIQR includes 21 items that are answered on a 0-10 numerical scale in which higher scores indicate greater functional impairment. The FIQR assesses the impact of FM symptoms over the past 7 days. The questionnaire consists of items that cover three domains: physical impairment, overall impact, and symptom severity. These items inquire about various aspects such as pain, energy levels, stiffness, sleep quality, depression, memory problems, anxiety, sensitivity to touch, balance issues, and heightened sensitivity to noises, lights, smells, or temperatures. The total FIQR score is calculated by summing the scores of the three subscales, resulting in a range of 0 to 100. Higher scores indicate a greater level of impairment. The Spanish version of the FIQR has an excellent internal consistency (α = 0.91-0.95)

SECONDARY OUTCOMES:
The Patient Global Impression of Change (PGIC) and the Pain Specific Impression of Change (PSIC) | At 3-months follow-up
  This instrument is an indicator of meaningful clinical change in treatments for chronic pain. The PGIC is one item (on a 7-point numerical scale, from 1 = 'Much better' to 7 = 'Much worse') referred to the participants' perception of global improvement due to treatment. It has undergone validation in the context of psychologically-based treatments for chronic pain. Additionally, the PSIC evaluates (also on a 7-point Likert scale) changes in specific domains, including physical and social functioning, work-related activities, mood, and pain. Both the PGIC & PSIC scales will be completed by participants assigned to STANZA and FM-ST treatments.
The Depression Anxiety Stress Scales-21 (DASS-21) | Through study completion, an average of 6 months
  It discriminates between features of depression, anxiety and stress in clinical and non-clinical samples. Responders are required to indicate the presence of several symptoms over the previous week. Each item is scored from 0 (´Did not apply to me at all over the last week') to 3 ('applied to me very much or most of the time over the past week'). There are 7 items on each of the three subscales: depression, anxiety and stress. Therefore, total scores in each scale can range from 0 to 21, with higher scores indicating more severe levels of depression, anxiety and stress. The Spanish version has excellent psychometric properties.
The Multidimensional Inventory of Subjective Cognitive Impairment (MISCI) | Through study completion, an average of 6 months
  It is a 10-item self-report measure of subjective cognitive dysfunction in FM during the last week. Each item is scored from 1 ('Not at all/Never') to 5 ('Very much/Always') and the total score ranges from 10 to 50. Lower scores indicate higher cognitive dysfunction. The MISCI was developed through classical test theory and item response theory from cognitive functioning item banks developed within the Patient Reported Outcomes Measurement Information System (PROMIS). The Spanish version of the MISCI has excellent internal reliability (α = 0.91)
The Pain Catastrophising Scale (PCS) | Through study completion, an average of 6 months
  Scale of 13 items comprising three dimensions: rumination over pain, magnification of pain and helplessness in the face of pain symptoms. The PCS total score and subscale scores are computed as the sum of ratings for each item.
  This study uses the total score, which can vary from 0 to 52 with higher scores indicating greater pain catastrophising.

OTHER OUTCOMES:
Psychological Inflexibility in Pain Scale (PIPS) | Through study completion, an average of 6 months.
  12-item scale that assesses psychological inflexibility in patients with pain and includes two factors: avoidance and cognitive fusion with pain. For this study, only the total score is used; it ranges from 12 to 84, with higher scores indicating higher level of psychological inflexibility.
EuroQoL (EQ-5D-5L) | Through study completion, an average of 6 months
  Instrument for evaluating health-related quality of life. The EQ-5D-5L scores will be used to calculate the Quality-Adjusted Life Years (QALYs) for the cost-utility analysis
Credibility/Expectancy questionnaire (CEQ) | Baseline
  6-item questionnaire for measuring treatment expectancy and credibility for use in clinical outcome studies. Each item is rated from 0 to 10, with higher scores indicating better expectancy.
Client Service Receipt Inventory (CSRI) | Through study completion, an average of 6 months
  The version used in this study is designed to retrospectively collect information on the use of health and social services during the previous six months. This instrument does not provide total or sub-scale scores, only collects information about use of services and medication consumption.
Adverse effects of therapies | Through study completion, an average of 6 months
  Qualitative ad hoc measure to check the presence of negative effects of the therapies
Socio-demographic and clinical questionnaire | Baseline
  Gender, date of birth, marital status, living arrangements, educational level, employment status, and years lived with fibromyalgia
Immune biomarkers | Baseline and 3-months follow-up
  Serum levels of IL-4, IL-6, CXCL8, IL-10, IL-17A, brain-derived neurotrophic factor (BDNF), and high sensitivity C-reactive protein (hs-CRP)
Hair cortisol and cortisone, serum cortisol, corticosteroid-binding globulin (CBG) and vitamin D. | Baseline and 3-months follow-up
  Biomarkers associated with HPA-axis functioning
Polymorphisms in the FKBP5 gene | Baseline
  Genetic variants of the FKBP5 gene. Five proposed SNP polymorphisms in the FKBP5 gene [rs3800373 (SNP1), rs9296158 (SNP2), rs1360780 (SNP3), rs9470080 (SNP4) and rs4713916 (SNP5)].

CONTACTS AND LOCATIONS:
Overall Officials: Juan V Luciano, PhD, Principal Investigator — Universitat Autònoma de Barcelona (UAB) & FSJD
Locations (2):
- Spain (2):
  - Parc Sanitari Sant Joan de Déu (PSSJD), Sant Boi de Llobregat, Barcelona
  - Hospital Vall d'Hebrón, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Catella S, Gendreau RM, Kraus AC, Vega N, Rosenbluth MJ, Soefje S, Malhotra S, Luciano JV, McCracken LM, Williams DA, Arnold LM. Self-guided digital acceptance and commitment therapy for fibromyalgia management: results of a randomized, active-controlled, phase II pilot clinical trial. J Behav Med. 2024 Feb;47(1):27-42. doi: 10.1007/s10865-023-00429-3. Epub 2023 Jun 29. PMID 37382794